CLINICAL TRIAL: NCT05883046
Title: The Acute Effects of Pre-Exercise Isolated and Combined Caffeine and Sodium Bicarbonate Consumption on Isometric Mid-thigh Pull Performance: A Placebo-Controlled Study
Brief Title: The Acute Effects of Combined Caffeine and Sodium Bicarbonate Consumption on Isometric Mid-thigh Pull
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Izzet Kirkaya, Associate Professor, Bozok University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BozokU-SBF-IK-01
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Athletes
Keywords: Caffeine; Sodium Bicarbonate; Isometric Contraction; Performance-Enhancing Substances
MeSH Terms: interventions — Performance-Enhancing Substances; BaseLine dental cement

STUDY DESIGN:
Intervention Model Description: subjects participated under 5 crossover conditions: control (without supplement) (Con), placebo (maltodextrin) (Pla), caffeine (Caf), sodium bicarbonate (NaHCO3) and caffeine+sodium bicarbonate (Caf+NaHCO3). The control measurement was made as a baseline measurement without supplementation.
Who Masked: Participant, Investigator
Masking Description: Supplement preparation, as well as the provision and management of blind conditions for both participants and investigators, were performed by a researcher (Celil KAÇOĞLU) who did not participate in the strength measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Baseline (Other): The control measurement was made as a baseline measurement without supplementation
  Interventions: Other: Baseline (Control)
- Placebo (Placebo Comparator): During Placebo conditions, participants consumed 20gr of maltodextrin (European origin, Alfasol®, Kimbiotek, Turkey).
  Interventions: Other: Placebo
- Caffeine (Experimental): For Caffeine conditions, participants consumed 6 mg/kg of caffeine, obtained from dosing the content of 200 mg capsules (Nature's Supreme® Caffeine)
  Interventions: Other: Performance-Enhancing Substances
- NaHCO3 (Experimental): As for NaHCO3 conditions, participants consumed 0.3 g/kg of sodium bicarbonate (Alfasol®, Kimbiotek, Turkey) dissolved in water
  Interventions: Other: Performance-Enhancing Substances
- Combined (Experimental): For the combined condition, (Caf+NaHCO3), 6 mg/kg of caffeine and 0.3 g/kg of sodium bicarbonate per kilogram of body weight of participants were consumed, after being dissolved together in water
  Interventions: Other: Performance-Enhancing Substances

INTERVENTIONS:
Other: Performance-Enhancing Substances — All supplements were consumed 60 min before the isometric mid-thigh pull tests, to reach peak blood concentrations at evaluation time. Immediately after consumption, both Control and intervention participants rested in a quiet laboratory environment (Eskişehir Technical University, Laboratory of Human Athletic Performance), until the strength tests. Participants were previously informed verbally and in writing that they should abstain from caffeine consumption (any caffeine-containing beverages and foods, such as coffee or tea, energy drinks, cocoa and cocoa-containing foods, chocolate and chocolate-containing foods or caffeine-containing drugs) for at least 24 hours before
  Arms: Caffeine; Combined; NaHCO3
Other: Placebo — 20gr of maltodextrin (European origin, Alfasol®, Kimbiotek, Turkey)
  Arms: Placebo
Other: Baseline (Control) — No supplement conditions
  Arms: Baseline

SUMMARY:
The aim of this study was to investigate the effects of isolated and combined caffeine and sodium bicarbonate consumption on acute isometric mid-thigh pull (IMTP) strength, and verify whether they are cumulative, neutral or subtractive.

DETAILED DESCRIPTION:
Method: Nineteen Sport Sciences Faculty students (Age 23.6±1.6 years, height 171±9.4 cm, weight 64.3±9.6 kg, fat percentage 20.5±7.3 %, BMI 21.7±2.4 kg/m2) participated and completed the intervention. This study was designed as crossover, double-blind and placebo-controlled. Subjects participated under 5 crossover conditions: control (without supplement) (Con), placebo (Pla), caffeine (Caf), sodium bicarbonate (NaHCO3) and caffeine+sodium bicarbonate (Caf+NaHCO3). For Caf conditions, participants consumed 6 mg/kg of caffeine, obtained from dosing the content of 200 mg capsules. As for NaHCO3 conditions, participants consumed 0.3 g/kg of sodium bicarbonate dissolved in water. For the combined condition, (Caf+NaHCO3), intake was set at 6 mg of caffeine and 0.3 g of sodium bicarbonate per kilogram of body weight. All supplements were consumed 60 min before the tests. Two submaximal trials of IMTP were performed at increasing intensities for 5 seconds (approximately %40-60 and %60-80 of their individually perceived 1RM, respectively, with 60-second rest intervals).

ELIGIBILITY:
Inclusion Criteria:

* Being physically active and healthy
* Did not use ergogenic supplements in the last 3 months
* Did not consume high doses of caffeine (≤120-170 mg/d) were included in this study

Exclusion Criteria:

* Actively using supplements
* Did not perform maximal effort during performance tests
* Not using the supplements in the correct dose or vomiting after use

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-12 (Actual)

PRIMARY OUTCOMES:
Isometric Mid-Thigh Pull (IMTP) | immediately after the intervention
  to investigate the effects of isolated and combined caffeine and sodium bicarbonate consumption on acute isometric mid-thigh pull (IMTP) strength, and verify whether they are cumulative, neutral or subtractive

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sport Sciences Eskisehir Technical University, Eskişehir, Tepebasi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data presented in this study are available on website https://osf.io/r6uz2/ with Identifier: 10.17605/OSF.IO/R6UZ2
Supporting Information: Study Protocol, Analytic Code
URL: https://osf.io/r6uz2/